CLINICAL TRIAL: NCT05361629
Title: The Effect of the Combination of Excision and Intraoperative Steroid Administration in Idiopathic Granulomatous Mastitis
Brief Title: Idiopathic Granulomatous Mastitis Combination Therapy
Acronym: IGM-COMBO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Huseyin Ozgur Aytac, Assoc Prof, Baskent University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MF 22-02
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Idiopathic Granulomatous Mastitis
Keywords: Idiopathic granulomatous mastitis; Steroid injection; Topical steroid; Steroid injection to surgical cavity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NON-SURGERY GROUP (Active Comparator): Group 1: Patients whose serum cortisol level was observed before starting the treatment, who were injected with 40 mg of prednol at 4 weeks intervals for 3 months for each lesion. The total monthly dose will not exceed 120 mg, and the total 3-month dose will not exceed 200 mg. In this group of patients, the serum cortisol level should have reappeared on the 2nd or 3rd day following each intralesional administration. In this group of patients, low-dose oral prednol (<30 mg/day) and/or topical prednol cream can be applied twice a day during the treatment.
  Interventions: Procedure: Intralesional steroid administration
- SURGERY GROUP (Active Comparator): In patients included in Group 2, serum cortisol levels should have been observed before starting treatment. Then the patients should be operated and the mass(s) should be excised. Intraoperatively, not less than 40 mg of prednol should be injected into each mass cavity (it may vary according to the cavity diameter), and the amount applied to all cavities should not exceed 200 mg in total. The amount of prednol administered for each cavity should be recorded. In this group of patients, prednol may have been administered to the cavity walls (Group 2a) or inside the cavity (Group 2b). Serum cortisol levels should be seen in patients 7 to 10 days after the procedure.
  Group 2a: 4 Quadrants 40 mg predmol per cavity wall (for < 2cm lesion and an additional 20 mg for each additional 1 cm) Group 2b: 40 mg predmol into the cavity (for < 2 cm lesion and an additional 20 mg for each additional 1 cm)
  Interventions: Procedure: Intraoperative cavity steroid administration

INTERVENTIONS:
Procedure: Intralesional steroid administration — Treatment by administering steroids into the lesion
  Arms: NON-SURGERY GROUP
Procedure: Intraoperative cavity steroid administration — Treatment by administering steroids into the surgical cavity
  Arms: SURGERY GROUP

SUMMARY:
After breast cancer, diopathic Granulomatous Mastitis (IGM) is among the breast diseases that bother patients and clinicians the most. Countries with a coast to the Mediterranean, especially our country, are the most common geography of this disease. For this reason, a significant part of the important scientific publications about IGM in the last 3-4 decades are from the countries of this geography and mainly from our country. The paradigm of whether IGM should be treated medically or surgically is still a matter of debate. Today, effective treatment results can be achieved with medical treatments, and local drug applications are finding an increasing application area in order to reduce the systemic drug level due to the side effects often seen in this process. As in the centers dealing with breast diseases intensively in our country, patients are treated in our center both by systemic and local means.

Within the body of the Turkish Breast Diseases Federation, after the plans made with the employees of the leading breast centers of the International Breast Health Working Group International planned to start a recording study to observe the activity between, local treatment in the lesion without surgical treatment with systemic treatment in IGM treatment and local treatment together with surgical treatment.

DETAILED DESCRIPTION:
AIM:

Primary: The effect of the combination of excision and single dose intraoperative steroid administration to the cavity on the shortening of the recovery period in Idiopathic Granulomatous Mastitis.

Secondary: Comparison of the side effects and the relationship between the treatment method and the serum cortisol level in patients treated with intralesional steroid + low dose oral steroid and topical steroid

THE WORK PLAN:

A prospective registry study was designed to compare the effectiveness of the combination of intralesional steroid administration used in the treatment of IGM + low-dose oral steroid therapy used together with the combination of surgical excision and intraoperative intra-cavity steroid administration.

For this purpose, it was planned to observe treatment success rates, time to treatment, recurrence rates at the earliest 1 year follow-up, and side effects related to surgical oral steroid use in eligible IGM patients treated in two different treatment groups.

METHOD:

After clinical and radiological evaluation, histopathological examination will be performed from core biopsy samples taken under ultrasound guidance and tuberculosis (TB) PCR and microbiological culture evaluation will be performed in all patients to rule out specific granulomatous inflammation. Patients with granulmatous inflammation characterized by histopathologically noncaseating granulomas, TB PCR negative and without culture growth, who meet the inclusion criteria, will be recruited into one of the two main treatment arms, at the discretion of the treating centre. There will be no randomization in determining the method of treatment. The type of treatment will be chosen according to the facilities of the performing center, especially the availability of intermittent access to the hospital for non-surgical treatment, and the priority to be determined between the patient and the physician. Since the efficiency superiority between the two methods is not known, any one will not be prioritized and the choice of treatment method will be determined by the patient and the physician. Among these patients, in those with localized abscess type IGM, the abscess foci that are present at the stage of sampling for TB PCR, microbiology culture and histopathology evaluation will be completely aspirated before the treatment is started, and will be waited until the sample results are obtained.

Treatment arms:

Group 1 (NON-SURGERY GROUP): Intralesional steroid + Low dose oral steroid (<30 mg/day prednol) Group 2 (SURGERY GROUP): Excision + Intraoperative steroid injection

Group 1: Patients whose serum cortisol level was observed before starting the treatment, who were injected with 40 mg of prednol at 4 weeks intervals for 3 months for each lesion. The total monthly dose will not exceed 120 mg, and the total 3-month dose will not exceed 200 mg. In this group of patients, the serum cortisol level should have reappeared on the 2nd or 3rd day following each intralesional administration. In this group of patients, low-dose oral prednol (<30 mg/day) and/or topical prednol cream can be applied twice a day during the treatment.

In patients included in Group 2, serum cortisol levels should have been observed before starting treatment. Then the patients should be operated and the mass(s) should be excised. Intraoperatively, not less than 40 mg of prednol should be injected into each mass cavity (it may vary according to the cavity diameter), and the amount applied to all cavities should not exceed 200 mg in total. The amount of prednol administered for each cavity should be recorded. In this group of patients, prednol may have been administered to the cavity walls (Group 2a) or inside the cavity (Group 2b). Serum cortisol levels should be seen in patients 7 to 10 days after the procedure.

Group 2a: 4 Quadrants 40 mg predmol per cavity wall (for < 2 cm lesion and an additional 20 mg for each additional 1 cm) Group 2b: 40 mg predmol into the cavity (for < 2 cm lesion and an additional 20 mg for each additional 1 cm)

Monitoring parameters:

* Recovery rates
* Time to recovery
* Recurrence rates after one-year follow-up
* Complications / side effects due to surgery or oral steroid use
* Relationship between steroid administration method and serum cortisol level Recovery (remission) was defined as the complete disappearance of pre-treatment clinical and ultrasonographic mastitis findings for patients in Group 1, and completion of wound healing for patients in Group 2.

Relapse was defined as the clinical or ultrasonographic re-detection of the disease in the same breast in both groups, following remission, in a similar or different type to the pre-treatment. Any need for repetitive surgery in the surgical arm will also be considered a recurrence.

In case of relapse in patients in both groups, the continuation of treatment will be left to the choice of centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with IGM histopathologically
* Patients in groups A, B and C according to clinical classification
* Ultrasonographically; Patients with leaf-like hypoechoic type, localized abscess type, and localized hypoechoic mass type mastitis

Exclusion Criteria:

* Patients diagnosed with tumor after biopsy
* Those with TB PCR (+)
* Presence of clinically widespread abscess and cellulite (group D patients)
* Ultrasonographically; diffuse diffuse type
* Pregnancy
* Breastfeeding period

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2022-04-16 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The effect of excision and intraoperative steroid administration to the cavity in Idiopathic Granulomatous Mastitis. | one year
  The effect of the combination of excision and single dose intraoperative steroid administration to the cavity on outcome in Idiopathic Granulomatous Mastitis.

SECONDARY OUTCOMES:
Rate of side effects in patients who received intralesional steroid | one year
  Comparison of side effect rates in patients treated with intralesional steroids +/- low-dose oral steroids and/or topical steroids.
Correlation of treatment modality and serum cortisol levels. | one year
  Correlation of treatment modality and serum cortisol levels in patients treated with intralesional steroids +/- low-dose oral steroids and/or topical steroids.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgur Aytac, MD, Study Director — Baskent University
Locations (1):
- Baskent University Adana Teaching Hospital, Adana, Yuregir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hu T, Li S, Huang H, Huang H, Tan L, Chen Y, Deng H, Wu J, Zhu L, Zhang J, Su F, Chen K. Multicentre, randomised, open-label, non-inferiority trial comparing the effectiveness and safety of ductal lavage versus oral corticosteroids for idiopathic granulomatous mastitis: a study protocol. BMJ Open. 2020 Oct 10;10(10):e036643. doi: 10.1136/bmjopen-2019-036643. PMID 33039992
- [Result] Ma X, Min X, Yao C. Different Treatments for Granulomatous Lobular Mastitis: A Systematic Review and Meta-Analysis. Breast Care (Basel). 2020 Feb;15(1):60-66. doi: 10.1159/000501498. Epub 2019 Jul 10. PMID 32231499
- [Result] Zhou F, Liu L, Liu L, Yu L, Wang F, Xiang Y, Zheng C, Huang S, Cai H, Yu Z. Comparison of Conservative versus Surgical Treatment Protocols in Treating Idiopathic Granulomatous Mastitis: A Meta-Analysis. Breast Care (Basel). 2020 Aug;15(4):415-420. doi: 10.1159/000503602. Epub 2019 Oct 22. PMID 32982653
- [Result] Wang Y, Song J, Tu Y, Chen C, Sun S. Minimally invasive comprehensive treatment for granulomatous lobular mastitis. BMC Surg. 2020 Feb 22;20(1):34. doi: 10.1186/s12893-020-00696-w. PMID 32087717